CLINICAL TRIAL: NCT00785096
Title: Perception of Surgical Complications - Agreements Among Patients, Nurses and Physicians
Brief Title: How do Patients, Nurses and Physicians Perceive Negative Postoperative Events?
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Ksenija Slankamenac, MD PhD, University of Zurich
Other Study IDs: 30-2008
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2015-02

CONDITIONS: Healthy
Keywords: Perception, surgical complications, patients, nurses and physicians
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Patients: Patients who admit for a minor or major surgical intervention
  Interventions: Other: Questionnaire
- Nurses: Medical staff of the University Hospital of Zurich
  Interventions: Other: Questionnaire
- Physicians: Medical staff of the University Hospital of Zurich and other institutions
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire, complications, grading severity, visual analog scale

SUMMARY:
The purpose of this study is to assess how patients, nurses and physicians perceive negative events following surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 18 years
* Capacity to act and no legal guardian
* Patients with any underlying disease admitted to the Department of Visceral and Transplantation Surgery of the University Hospital of Zurich with planned minor or major visceral surgery
* German language as daily language.

Exclusion Criteria:

* Patients with cognitive difficulties and diseases, which may yield unreliable answers
* Patients unable to read and write

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who will admit for a minor or major surgical procedure Nurses from the University Hospital of Zurich Different physicians of the University Hospital of Zurich (surgeons, anesthesia, urologist ans ICU-care specialists)and other institutions.
Sampling Method: Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
To assess how patients, nurses and physicians perceive negative events following surgical procedures | August 2008- December 2009

SECONDARY OUTCOMES:
Association to the Clavien Dindo Classification | August 2008 - December 2009

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Visceral and Transplantation Surgery of the University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland